CLINICAL TRIAL: NCT00434772
Title: Glucagon in the Treatment of Hypoglycemia in Newborn Infants of Diabetic Mothers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: bisseliches-glucagon-ctil
Record Dates: First submitted 2007-02-11; First posted 2007-02-13 (Estimated); Last update posted 2009-05-28 (Estimated); Status verified 2009-05

CONDITIONS: Hypoglycemia
Keywords: hypoglycemia; glucagon; neonatal; gestational diabetes; insulin; glyburide
MeSH Terms: conditions — Hypoglycemia; Diabetes, Gestational; Insulin Resistance | interventions — Glucagon

INTERVENTIONS:
Drug: glucagon

SUMMARY:
Thesis Infants of diabetic mothers are at high risk to develop hypoglycemia after birth.

After birth, glucose and ketone bodies are the main substrates of brain energy. Under normal condition, the adrenergic response seen immediately after birth suppresses insulin release and stimulates glucagon secretion which enhances gluconeogenesis and ketogenesis.

An inversion of the insulin/glucagon ratio is seen soon after birth as a normal, physiologic phenomenon. Consequently, a post delivery glucose nadir is reached between 30 to 90 minutes after birth, followed by a spontaneous recovery before 3-4 hours of age.

In infants of diabetic mothers, this inversion of the ratio is postponed and a more profound and sustained hypoglycemia is seen.

Early feeding is of great importance to diminish the severity and incidence of hypoglycemia. But, if despite an appropriate calorie intake, low levels of sugar are seen, an intravenous infusion of glucose should be commenced. In case that IV glucose is not effective or can't be supplied immediately, intramuscular glucagon is a therapeutic alternative.

We hypothesize that a single intramuscular injection of glucagon together with the appropriate oral intake of nutrients is a safe and an effective alternative to the IV infusion of glucose alone in the treatment of hypoglycemia in term infants of diabetic mothers.

Methods Appropriately grown or large for date, term infants of insulin treated diabetic mothers, with no other known medical problems, are potential candidates for our study.

Hypoglycemia will be defined as serum glucose level lower than 45 mg%. Infants of diabetic mothers will arrive to the nursery and immediately receive early feeding before 30 minutes of life. At that time, glucose will be checked. If glucose level is lower than 45 mg%, treatment with IV glucose or IM glucagon will be initiated. Glucose will be checked every hour for 4 hours and then every 3 hours (before each meal) for the next 20 hours.

In case blood glucose level is lower than 20 mg% or falls below 45 mg% despite glucagon treatment, IV glucose will immediately be instituted.

Our aim is to check that IM Glucagon is as good as IV glucose in the treatment of hypoglycemia in infants of diabetic mothers. We will compare glucose levels after treatment with IV glucose and IM glucagon, the time till normalization of glucose and full feeding is achieved and the number of hospitalization days in both groups.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic hypoglycemia
* infant of insulin treated diabetic mother
* AGA or LGA
* no other known medical problems

Exclusion Criteria:

* concurrent medical problems
* symptomatic hypoglycemia
* glucose under 20 mg%

Max Age: 48 Hours | Sex: All
Age Groups: Child
Dates: Start 2007-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
glucose

SECONDARY OUTCOMES:
hospitalisation days

CONTACTS AND LOCATIONS:
Overall Officials: Bisseliches Myriam, MD, Principal Investigator — Shaare Zedek Medical Center - Jerusalem - Israel
Locations (1):
- Share Zedek Medical Center, Jerusalem, Israel